CLINICAL TRIAL: NCT06797037
Title: Proof of Concept to Assess the Feasibility of a Decentralised Pathway Coordinated by the Advanced Practice Nurse for Patients Receiving Oral Treatment for Cancer or Malignant Haemopathy (ACCELER PLATFORM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24GENE18
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Solid Cancer; Haematological Malignancies
Keywords: Retroceded oral chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with solid cancer or haematological malignancies and requiring oral chemotherapy (Other)
  Interventions: Other: Decentralised Pathway Coordinated by the Advanced Practice Nurse

INTERVENTIONS:
Other: Decentralised Pathway Coordinated by the Advanced Practice Nurse — For each patient enrolled in the study: a decentralised treatment delivery route will be organised. To achieve this, two visits will be planned by the investigating centre's Advanced Practice Nurse (APN) and carried out at the patient's home by a service-providing nurse. During these visits, the APN will take the patient's vital signs before handing over the treatment.
  In addition, for the purposes of the study, during the 2nd visit the patient will be asked to complete a satisfaction questionnaire.

SUMMARY:
This is an open-label, single-centre, category 2 "Jardé Law" proof-of-concept study designed to demonstrate the feasibility of a decentralised care pathway for patients with cancer or haematological malignancies receiving oral treatment.

The study will be conducted on a population of 33 patients.

In current practice, patients with certain solid cancers or haematological malignancies may be prescribed oral chemotherapy on a retroceded basis. In these cases, the oncologist (coordinating investigator) sees the patient for a consultation every 3 cycles to prescribe/renew the treatment for approximately 3 months. Every month, the patient returns to the centre to have the treatment dispensed by the hospital pharmacy. No medical consultation is associated with this visit.

In this study, it is proposed to decentralise the delivery of treatment to these patients by introducing two visits to the patient's home by a service-providing nurse.

The decentralised patient pathway will be organised and monitored by the Advanced Practice Nurse (APN) at the investigating centre, who will be responsible in particular for coordination with the service-providing nurse and the hospital pharmacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18.
2. A patient with solid cancer or haematological malignancy receiving oral retroceded therapy as part of standard management.
3. Patient with a performance index (ECOG): 0-2.
4. Patient contactable by telephone for follow-up by the Advanced Practice Nurse.
5. Patient willing to make two home visits within 6 months of inclusion.

Exclusion Criteria:

1. Pregnant or breast-feeding patient.
2. Any psychological, family, geographical or social condition which, in the judgement of the oncologist, could potentially prevent the collection of informed consent or hinder compliance with the study protocol.
3. Patients deprived of their liberty by administrative or legal decision, or patients under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-05-19 (Estimated); Study Completion 2027-05-19 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was defined as the feasibility of decentralisation. | 7 months for each patient
  Feasibility is a composite criterion, defined according to two dimensions: exhaustive collection of clinical data and logistical feasibility. For a patient, decentralisation will be considered feasible if success is observed for both dimensions.

SECONDARY OUTCOMES:
Patient adherence to decentralised management. | 7 months for each patient
  This will be measured by the acceptance rate of trial participants compared with the number of proposals made.
Patient satisfaction with decentralised management. | 7 months for each patient
  This will be evaluated according to different components using a likert scale. Patients will be asked 10 questions to assess their satisfaction. There will be 5 possible answers ranging from 'completely agree' to 'completely disagree'.
Time taken to collect data from home to site. | 7 months for each patient
  This will be defined as the time between the date of the home visit and the date on which the data is 'uploaded' into the investigating centre's computerised patient record.
The rate of patients for whom the data interface well with the site's electronic patient record. | 7 months for each patient
  This is defined as the ratio of the number of patients for whom the data has been 'uploaded' into the electronic patient record to the total number of patients.
The operation of the outsourced computerised patient file tool (MHCare). | 7 months for each patient
  This will be assessed at each visit by the rate of patients for whom the tool worked well.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France